CLINICAL TRIAL: NCT03238027
Title: A Phase 1, Open-Label, Dose Escalation Trial to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Activity of SNDX-6352 Monotherapy and SNDX-6352 in Combination With Durvalumab in Patients With Unresectable, Recurrent, Locally-Advanced, or Metastatic Solid Tumors
Brief Title: A Phase 1 Study to Investigate Axatilimab Alone or in Combination With Durvalumab in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SNDX-6352-0502
Record Dates: First submitted 2017-06-30; First posted 2017-08-03 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Solid Tumor; Metastatic Tumor; Locally Advanced Malignant Neoplasm; Unresectable Malignant Neoplasm
Keywords: SNDX-6352; CSF-1R inhibitor; Colony Stimulating factor 1 receptor inhibitor; Solid Tumor; Recurrent locally advanced tumor; unresectable solid tumor; Metastatic tumor; durvalumab
MeSH Terms: conditions — Neoplasm Metastasis | interventions — axatilimab; durvalumab

STUDY DESIGN:
Intervention Model Description: Initially in both phases, 3 patients will receive axatilimab at 1 mg/kg IV on C1D1 and again on C1D15 of a 28-day cycle. Phase 1b only will also receive a fixed dose of 1500mg durvalumab IV on C1D1. If no DLTs are noted, 3 more patients will be treated at the next higher dose level (3 mg/kg). If 1 DLT is observed in 1 of 3 patients, 3 more patients will be treated at that starting dose level (1 mg/kg). If 2 or more DLTs are observed in 3-6 patients at the starting dose, the study will be terminated, or a lower dose will be considered. If the safety profile is acceptable, escalation to axatilimab doses of 3, 6 and 10mg/kg are planned for the 1a and for the 1b, doses of 3 and 6 mg/kg of axatilimab in combination with a fixed dose of 1500mg of durvalumab are planned. The MTD will be considered to have been exceeded if 2 or more patients in a dose group experience a DLT; in this case, the next lower dose group which has been evaluated will be considered as the MTD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Ph1a D1: 1 mg/kg Axatilimab (Experimental): Three (3) patients receive starting dose of 1 mg/kg of axatilimab and are followed for possible DLTs. If one DLT is observed in 1 of 3 patients, an additional 3 patients will be enrolled at this dose level. If no DLTs are noted in any of the 3 patients, next dosing arm will commence following review by Scientific Review Committee.
  Interventions: Drug: Axatilimab
- Ph1a D2: 3 mg/kg Axatilimab (Experimental): Three (3) patients receive next higher dose of 3 mg/kg of axatilimab and are followed for possible DLTs. If one DLT is observed in 1 of 3 patients, an additional 3 patients will be enrolled at this dose level. If no DLTs are noted in any of the 3 patients, next dosing arm will commence following review by Scientific Review Committee.
  Interventions: Drug: Axatilimab
- Ph1a D3: 6 mg/kg Axatilimab (Experimental): Three (3) patients receive next higher dose of 6 mg/kg of axatilimab and are followed for possible DLTs. If one DLT is observed in 1 of 3 patients, an additional 3 patients will be enrolled at this dose level. If no DLTs are noted in any of the 3 patients, next dosing arm will commence following review by Scientific Review Committee.
  Interventions: Drug: Axatilimab
- Ph1a D4: 10 mg/kg Axatilimab (Experimental): Three (3) patients receive next higher dose of 10 mg/kg of axatilimab and are followed for possible DLTs. If one DLT is observed in 1 of 3 patients, an additional 3 patients will be enrolled at this dose level. If no DLTs are noted in any of the 3 patients, next dosing arm will commence following review by Scientific Review Committee.
  Interventions: Drug: Axatilimab
- Ph1b D1: 1 mg/kg Axatilimab+1500 mg durvalumab (Experimental): Three (3) patients receive starting dose of 1 mg/kg of axatilimab every two weeks and 1500 mg durvalumab every four weeks and are followed for possible DLTs. If one DLT is observed in 1 of 3 patients, an additional 3 patients will be enrolled at this dose level. If no DLTs are noted in any of the 3 patients, next dosing arm will commence following review by Scientific Review Committee. If 1 DLT is observed in 1 of 3 patients, then 3 additional patients will be treated at the 1 mg/kg axatilimab dose level; if none of the 3 additional patients experience a DLT (i.e. 1 of 6), the dose will be escalated to an intermediate dose of 2 mg/kg. Escalation from 2 mg/kg to 3 mg/kg will follow the general dose escalation rules described above for both study phases.
  Interventions: Drug: Axatilimab; Drug: Durvalumab
- Ph1b D2: 3 mg/kg Axatilimab+1500 mg durvalumab (Experimental): Three (3) patients receive next higher dose of 3 mg/kg of axatilimab every two weeks and 1500 mg durvalumab every four weeks and are followed for possible DLTs. For cohorts with doses ≥3 mg/kg, a sentinel recruitment approach will be utilized. Initially 1 patient in each cohort will be treated with the combination therapy and safety will be evaluated by SRC at Cycle 1, Day 8; if no safety concerns are identified, the next 2 patients can be treated in that cohort. If one DLT is observed in 1 of 3 patients, an additional 3 patients will be enrolled at this dose level. If no DLTs are noted in any of the 3 patients, next dosing arm will commence following review by Scientific Review Committee.
  Interventions: Drug: Axatilimab; Drug: Durvalumab
- Ph1b D3: 6 mg/kg Axatilimab+1500 mg durvalumab (Experimental): Three (3) patients receive next higher dose of 6 mg/kg of axatilimab every two weeks and 1500 mg durvalumab every four weeks and are followed for possible DLTs. For cohorts with doses ≥3 mg/kg, a sentinel recruitment approach will be utilized. Initially 1 patient in each cohort will be treated with the combination therapy and safety will be evaluated by SRC at Cycle 1, Day 8; if no safety concerns are identified, the next 2 patients can be treated in that cohort. If one DLT is observed in 1 of 3 patients, an additional 3 patients will be enrolled at this dose level. If no DLTs are noted in any of the 3 patients, next dosing arm will commence following review by Scientific Review Committee.
  Interventions: Drug: Axatilimab; Drug: Durvalumab

INTERVENTIONS:
Drug: Axatilimab — Humanized IgG4 mAb that blocks colony stimulating factor 1 receptor (CSF-1R)
  Other Names: SNDX-6352
Drug: Durvalumab — Durvalumab (MEDI4736) is a humanized IgG1 kappa mAb that blocks the interaction of PD-L1 with PD-1 CD80 (B7.1) molecules
  Other Names: MEDI4736
  Arms: Ph1b D1: 1 mg/kg Axatilimab+1500 mg durvalumab; Ph1b D2: 3 mg/kg Axatilimab+1500 mg durvalumab; Ph1b D3: 6 mg/kg Axatilimab+1500 mg durvalumab

SUMMARY:
A Phase 1 dose escalation study to determine if axatilimab as monotherapy and axatilimab in combination with a fixed dose of durvalumab will be sufficiently safe and well-tolerated at biologically active doses to warrant further investigation in patients with solid tumors.

DETAILED DESCRIPTION:
This is an open label, multi-center Phase 1 study consisting of Phase 1a and Phase 1b. The study will evaluate axatilimab monotherapy (in Phase 1a) and axatilimab combined with durvalumab (in Phase 1b) in patients with advanced solid tumors which must have progressed following prior treatment and have no standard therapy alternatives left (i.e., patients must not be candidates for regimens known to provide clinical benefit). The primary objective will be to determine the MTD and/or RP2D of axatilimab as monotherapy (Phase 1a) and in combination with durvalumab (Phase 1b) as evaluated by the incidence of AEs that are defined as DLTs. In both study phases, a standard "3+3" dose escalation schema will be used to determine an MTD with 3-6 evaluable patients enrolled per dose level. The RP2D will be determined based on data from the dose escalation patients as reviewed by the Safety Review Committee (SRC; comprised of investigators and the Sponsor).

ELIGIBILITY:
INCLUSION CRITERIA:

Inclusion Criteria for Phase 1a and Phase 1b

Patients meeting all of the following criteria are considered eligible to participate in the study:

1. Signed written informed consent form (ICF).
2. Male or female patients aged ≥18 years.
3. Patients with histopathologically confirmed unresectable, recurrent, locally advanced, or metastatic solid tumors, with evaluable disease and must have progressed following prior treatment and have no standard therapy alternatives left (i.e., patients must not be candidates for regimens known to provide clinical benefit).
4. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1 at the study enrollment.
5. Has adequate organ and bone marrow function within 21 days before enrollment as defined below:

   a. Hematological laboratory values: i. Absolute Neutrophil Count (ANC) ≥1.5 × 10^9/L ii. Platelets ≥100 × 10^9/L iii. Hemoglobin ≥9 g/dL b. Renal laboratory values: i. Creatinine ≤1.5 times the Upper Limit of Normal (ULN) OR ii. Measured or calculated (per institutional standard) creatinine clearance (CrCl) ≥60 mL/min according to the Cockcroft-Gault formula or measured 24-hour creatinine clearance (or local institutional standard measure) for patient with creatinine level > 1.5 times institutional ULN.

   iii. Glomerular filtration rate may be used instead of creatinine or CrCl. c. Hepatic laboratory values: i. Total bilirubin ≤1.5 times ULN or ii. Direct bilirubin ≤ULN for patients with total bilirubin >1.5 times ULN iii. AST and ALT ≤2.5 times ULN d. Creatine kinase ≤ ULN
6. Experienced resolution of toxic effect(s) of the most recent prior anti-cancer therapy to Grade ≤1 (except alopecia) per NCI CTCAE v5.0 If a patient underwent major surgery or radiation therapy of >30 Gray, the patient must have recovered from the toxicity and/or complications from the intervention.

   Note: Patients with ≤ Grade 2 neuropathy or ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study.
7. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
   * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
8. Female patients of childbearing potential who are not abstinent and intend to be sexually active with a nonsterilized male partner must use at least 1 highly effective method of contraception (Table 11) from the time of screening throughout the total duration of the study drug treatment and 90 days after the last dose of study drug. Non-sterilized male partners of a female patient of childbearing potential must use male condom plus spermicide throughout this period. Cessation of birth control after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Female patients should also refrain from breastfeeding throughout this period.
9. Non-sterilized male patients who are not abstinent and intend to be sexually active with a female partner of childbearing potential must use a male condom plus spermicide from the time of screening throughout the total duration of the study drug treatment and 90 days after the last dose of study drug. However, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Male patients should refrain from sperm donation throughout this period.
10. Must have a life expectancy of at least 12 weeks.

Additional Inclusion Criteria for Phase 1b 11. Body weight > 30 kg 12. No prior exposure to immune-mediated therapy including, but not limited to, other anti CTLA-4, anti-PD-1, anti-PD-L1, and anti-PD-L2 antibodies, excluding therapeutic anticancer vaccines.

EXCLUSION CRITERIA:

Exclusion Criteria for Phase 1a and Phase 1b

Patients meeting any of the following criteria are not eligible for study participation:

1. Diagnosis of immunodeficiency or receiving systemic corticosteroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of study drug.

   a. Exceptions: 1) The use of physiologic doses of corticosteroids (i.e., ≤10 mg per day of equivalent prednisone) is allowed; 2) Steroids with no or minimal systemic effect (topical, inhalation) are allowed; 3) Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment; (4) Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
2. Previously treated with a CSF-1, CSF-1R, and/or IL-34-blocking agents
3. Psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
4. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the patient's best interest to participate, in the opinion of the treating Investigator, including, but not limited to:

   1. Active or prior documented autoimmune or inflammatory disorders (see Appendix 3 for complete list).
   2. History of active primary immunodeficiency
   3. Known active or latent tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice).
   4. Myocardial infarction or arterial thromboembolic events within 6 months prior to enrollment or severe or unstable angina, New York Heart Association (NYHA) (see Appendix 2) Class III or IV disease, or a QTc interval > 470 msec. History of QTc prolongation, ventricular fibrillation, ventricular tachycardia or Torsades de Pointes (TdP).
   5. Symptomatic congestive heart failure, cardiac arrhythmia, uncontrolled hypertension or diabetes mellitus.
   6. Active infection requiring systemic therapy.
   7. Interstitial lung disease
   8. Serious chronic gastrointestinal conditions associated with diarrhea
   9. Has untreated central nervous system (CNS) metastases and/or carcinomatous meningitis identified either on the baseline brain imaging (please see Appendix A (RECIST)) for details on the imaging modality) obtained during the screening period or identified prior to signing the ICF. Patients whose brain metastases have been treated may participate provided they show radiographic stability (defined as 2 brain images, both of which are obtained after treatment to the brain metastases. These imaging scans should both be obtained at least four weeks apart and show no evidence of intracranial progression). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either, without the use of steroids, or are stable on a steroid dose of ≤10 mg/day of prednisone or its equivalent for at least 14 days prior to the start of treatment. Brain metastases will not be recorded as RECIST Target Lesions at baseline.
5. Received a live attenuated vaccine within 30 days of the first dose of study drug.

   Note: Patients, if enrolled, should not receive live vaccine whilst receiving study drug and up to 30 days after the last dose of study drug.
6. Administration of colony stimulating factors (including granulocyte-colony stimulating factor [G-CSF], granulocyte macrophage-colony stimulating factor [GM-CSF], or recombinant erythropoietin) within 4 weeks prior to the first dose of study drug treatment.
7. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
8. Received chemotherapy, anti-cancer mAb, targeted small molecule or other systemic anti-cancer therapy within 4 weeks of the first dose of study drug. However, patients receiving conventional and investigational small molecule targeted therapies that are not expected to have delayed toxicities may enter the study 5 half-lives or 28 days after the last dose of the compound, whichever is shorter.
9. Currently receiving treatment with any other agent listed on the prohibited medication list.
10. Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
11. Known active hepatitis B (e.g., hepatitis B surface antigen-reactive) or hepatitis C (e.g., hepatitis C virus ribonucleic acid [qualitative]). Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBc Ab] and absence of HBsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
12. Known alcohol or drug abuse.
13. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
14. Legal incapacity or limited legal capacity.
15. Evidence of muscle disorders or muscle injury that are known to cause serum creatine kinase (CK) elevation
16. Current pneumonitis or has a history of (non-infectious) pneumonitis that required steroids
17. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
18. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study drug. Note: Local surgery of isolated lesions for palliative intent is acceptable.
19. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks or palliative radiation therapy within 2 weeks of the first dose of study drug
20. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of study drug

    Additional Exclusion Criteria for Phase 1b
21. History of allogenic organ transplantation.
22. Patients who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Phase 1a: Determination of any Dose limiting toxicities (DLT)s of Axatilimab | Approximately 9 months (from first dose to 90-day follow-up post-last dose)
  All patients treated with axatilimab across all treatment arms (dosing levels) will have safety assessed in order to determine any dose-limiting toxicities (DLT)s.
Phase 1a: Determination of Maximum tolerable dose (MTD) of Axatilimab | Approximately 9 months (from first dose to 90-day follow-up post-last dose)
  All patients treated with axatilimab across all treatment arms (dosing levels) will have safety assessed in order to determine the MTD.
Phase 1a: Determination of Recommended Phase 2 dose (RP2D) of Axatilimab | Approximately 9 months (from first dose to 90-day follow-up post-last dose)
  All patients treated with axatilimab across all treatment arms (dosing levels) will have safety assessed in order to determine the RP2D.
Phase 1b: Determination of any Dose limiting toxicities (DLT)s of Axatilimab when given in combination with a fixed dose of durvalumab | Approximately 9 months (from first dose to 90-day follow-up post-last dose)
  All patients treated with axatilimab in combination with a fixed dose of durvalumab across all treatment arms (dosing levels) will have safety assessed in order to determine any dose-limiting toxicities (DLT)s.
Phase 1b: Determination of Maximum tolerable dose (MTD) of Axatilimab when given in combination with a fixed dose of durvalumab | Approximately 9 months (from first dose to 90-day follow-up post-last dose)
  All patients treated with axatilimab in combination with a fixed dose of durvalumab across all treatment arms (dosing levels) will have safety assessed in order to determine the MTD.
Phase 1b: Determination of Recommended Phase 2 dose (RP2D) of Axatilimab when given in combination with a fixed dose of durvalumab | Approximately 9 months (from first dose to 90-day follow-up post-last dose)
  All patients treated with axatilimab in combination with a fixed dose of durvalumab across all treatment arms (dosing levels) will have safety assessed in order to determine the RP2D.

SECONDARY OUTCOMES:
Phase 1a: PK endpoint of Cmax (maximum observed concentration) for Axatilimab as dose levels increase across different treatment groups. | Approximately 6 months (from first dose to End of Treatment visit)
  Cmax for SDNX-6352 for axatilimab will be computed.
Phase 1a: PK endpoint of AUC (area under the curve) for Axatilimab as dose levels increase across different treatment groups. | Approximately 6 months (from first dose to End of Treatment visit)
  AUC for SDNX-6352 for axatilimab will be computed.
Phase 1a: PK endpoint of Tmax (time to reach maximum observed concentration) for Axatilimab as dose levels increase across different treatment groups. | Approximately 6 months (from first dose to End of Treatment visit)
  Tmax for SDNX-6352 for axatilimab will be computed.
Phase 1a: PK endpoint of T1/2 (apparent terminal elimination half life)) for Axatilimab as dose levels increase across different treatment groups. | Approximately 6 months (from first dose to End of Treatment visit)
  T1/2 for SDNX-6352 for axatilimab will be computed.
Phase 1a: Evaluation of preliminary anti-tumor activity of Axatilimab on solid tumors | Approximately 9 months (from baseline scan to 90-day follow-up post-last dose)
  To determine if the size and number of target lesions changes in response to treatment with axatilimab by analyzing CT-Scans/MRIs per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) and irRECIST.
Phase 1a: Effect of Axatilimab on CSF-1 and IL-34 | Approximately 6 months (from first dose to End of Treatment visit)
  To assess change from Baseline in plasma CSF-1 and IL-34 following IV administration
Phase 1a: Evaluate the immunogenicity of Axatilimab | Approximately 6 months (from first dose to End of Treatment visit)
  To assess the immunogenicity of axatilimab as measured by presence of anti-drug antibodies (ADA)
Phase 1b: PK endpoint of Cmax (maximum observed concentration) for Axatilimab when given in combination with a fixed dose of durvalumab as dose levels increase across different treatment groups. | Approximately 6 months (from first dose to End of Treatment visit)
  Cmax for axatilimab will be computed.
Phase 1b: PK endpoint of AUC (area under the curve) for Axatilimab when given in combination with a fixed dose of durvalumab as dose levels increase across different treatment groups. | Approximately 6 months (from first dose to End of Treatment visit)
  AUC for axatilimab will be computed.
Phase 1b: PK endpoint of Tmax (time to reach maximum observed concentration) for Axatilimab when given in combination with a fixed dose of durvalumab as dose levels increase across different treatment groups. | Approximately 6 months (from first dose to End of Treatment visit)
  Tmax for axatilimab will be computed.
Phase 1b: PK endpoint of T1/2 (apparent terminal elimination half-life)) for Axatilimab when given in combination with a fixed dose of durvalumab as dose levels increase across different treatment groups. | Approximately 6 months (from first dose to End of Treatment visit)
  T1/2 for axatilimab will be computed.
Phase 1b: PK endpoint of Cmax (maximum observed concentration) for durvalumab when given in combination with Axatilimab as dose levels increase across different treatment groups. | Approximately 6 months (from first dose to End of Treatment visit)
  Cmax for durvalumab will be computed.
Phase 1b: PK endpoint of AUC (area under the curve) for durvalumab when given in combination with Axatilimab as dose levels increase across different treatment groups. | Approximately 6 months (from first dose to End of Treatment visit)
  AUC for durvalumab will be computed.
Phase 1b: PK endpoint of Tmax (time to reach maximum observed concentration) for durvalumab when given in combination with Axatilimab as dose levels increase across different treatment groups. | Approximately 6 months (from first dose to End of Treatment visit)
  Tmax for durvalumab will be computed.
Phase 1b: PK endpoint of T1/2 (apparent terminal elimination half-life) for durvalumab when given in combination with Axatilimab as dose levels increase across different treatment groups. | Approximately 6 months (from first dose to End of Treatment visit)
  T1/2 for durvalumab will be computed.
Phase 1b: Evaluation of preliminary anti-tumor activity of Axatilimab when given in combination with a fixed dose of durvalumab on solid tumors. | Approximately 9 months (from baseline scan to 90-day follow-up post-last dose)
  To determine if the size and number of target lesions changes in response to treatment with axatilimab by analyzing CT-Scans/MRIs per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) and irRECIST.
Phase 1b: Effect of Axatilimab on CSF-1 and IL-34 | Approximately 6 months (from first dose to End of Treatment visit)
  To assess change from Baseline in plasma CSF-1 and IL-34 following IV administration
Phase 1b: Evaluation of the immunogenicity of Axatilimab | Approximately 6 months (from first dose to End of Treatment visit)
  To assess the immunogenicity of axatilimab as measured by presence of anti-drug antibodies (ADA)
Phase 1b: Evaluation of the immunogenicity of durvalumab | Approximately 6 months (from first dose to End of Treatment visit)
  To assess the immunogenicity of durvalumab as measured by presence of anti-drug antibodies (ADA)

OTHER OUTCOMES:
Phase 1a: Effect of Axatilimab on CSF-1 receptor occupancy | Approximately 6 months (from first dose to End of Treatment visit)
  To evaluate the change from Baseline in CSF-1 receptor occupancy (RO)
Phase 1a: Exploration of relationship between candidate biomarker results and anti-tumor activity of Axatilimab | Approximately 6 months (from first dose to End of Treatment visit)
  To investigate the relationship between candidate biomarkers (e.g., CSF-1, IL-34) and anti-tumor activity of axatilimab
Phase 1a: Exploration of relationship between additional biomarkers and anti-tumor activity of Axatilimab | Approximately 6 months (from first dose to End of Treatment visit)
  To investigate the relationship between other biomarkers (e.g., tumor infiltrating lymphocytes, PD-L1, PD-1, PD-L2, circulating classical and non-classical CD-16 monocytes in blood) and anti-tumor activity of axatilimab
Phase 1a: Characterization of relationship in change from baseline in CSF-1, IL-34, etc. with Axatilimab administered intravenously. | Approximately 6 months (from first dose to End of Treatment visit)
  To characterize the relationship in change from baseline in plasma colony stimulating factor-1 [CSF-1] interleukin-34 [IL-34]), and IFN-gamma, IL-1beta, IL-2, IL-4, IL-5, IL-6, CXCL8/IL-8, IL-10, IL-12 (p70), IL-13, TNF-alpha, CD204/206 and sCD163 with systemic PK of axatilimab administered intravenously.
Phase 1b: Characterization of the PD profile of Axatilimab and durvalumab when given in combination. | Approximately 6 months (from first dose to End of Treatment visit)
  To characterize the pharmacodynamic (PD) profile of axatilimab and durvalumab when given in combination in patients with advanced solid tumors.
Phase 1b:Effect of Axatilimab when given in combination with a fixed dose of durvalumab on CSF-1 receptor occupancy. | Approximately 6 months (from first dose to End of Treatment visit)
  To evaluate the change from Baseline in CSF-1 receptor occupancy (RO).
Phase 1b: Exploration of relationship between candidate biomarker results and anti-tumor activity of Axatilimab when given in combination with a fixed dose of durvalumab. | Approximately 6 months (from first dose to End of Treatment visit)
  To investigate the relationship between candidate biomarkers (e.g., CSF-1, IL-34) and anti-tumor activity of axatilimab when given in combination with a fixed dose of durvalumab.
Phase 1b: Exploration of relationship between additional biomarkers and anti-tumor activity of Axatilimab when given in combination with a fixed dose of durvalumab. | Approximately 6 months (from first dose to End of Treatment visit)
  To investigate the relationship between other biomarkers (e.g., tumor infiltrating lymphocytes, PD-L1, PD-1, PD-L2, circulating classical and non-classical CD-16 monocytes in blood) and anti-tumor activity of axatilimab when given in combination with a fixed dose of durvalumab.
Phase 1b: Characterization of relationship in change from baseline in CSF-1, IL-34, etc. with Axatilimab administered intravenously when given in combination with a fixed dose of durvalumab. | Approximately 6 months (from first dose to End of Treatment visit)
  To characterize the relationship in change from baseline in plasma colony stimulating factor-1 [CSF-1] interleukin-34 [IL-34]), and IFN-gamma, IL-1beta, IL-2, IL-4, IL-5, IL-6, CXCL8/IL-8, IL-10, IL-12 (p70), IL-13, TNF-alpha, CD204/206 and sCD163 with systemic PK of axatilimab administered intravenously when given in combination with a fixed dose of durvalumab.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Madigan, MD, Study Director — Syndax Pharmaceuticals
Locations (5):
- United States (5):
  - Honor Health, Scottsdale, Arizona
  - Johns Hopkins University, Baltimore, Maryland
  - Oregon Health and Science University, Portland, Oregon
  - NEXT Oncology, San Antonio, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No